CLINICAL TRIAL: NCT05649306
Title: Gender Related Coping and Survivorship for Genitourinary Cancers
Status: Recruiting | Type: Observational
Sponsor: Johns Hopkins University (Other)
Responsible Party: Sponsor
Other Study IDs: IRB00314755
Record Dates: First submitted 2022-12-01; First posted 2022-12-14 (Actual); Last update posted 2025-10-03 (Actual); Status verified 2025-10

CONDITIONS: Bladder Cancer
Keywords: Female; Adult; Genitourinary Cancers
MeSH Terms: conditions — Urinary Bladder Neoplasms; Urogenital Neoplasms | interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (4):
- Patients not receiving a cystectomy - Standard of Care Group: Patients will receive standard of care treatment. Patients will be asked to complete the Demoralization Scale II and Female Sexual Function Index at baseline, 1-month following treatment, 3-months following treatment, 6-months following treatment, and one-year following treatment.
  Interventions: Other: Questionnaires
- Patients not receiving a cystectomy - Additional Education Group: Patients will receive additional education with standard of care treatment. Patients will be asked to complete the Demoralization Scale II and Female Sexual Function Index at baseline, 1-month following treatment, 3-months following treatment, 6-months following treatment, and one-year following treatment. Patients will also be asked to complete an attendance diary documenting additional support services utilized. The Attendance Diary will be completed at 1-month following treatment, 3-months following treatment, 6-months following treatment, and one-year following treatment.
  Interventions: Other: Additional Education; Other: Attendance Diary
- Patients receiving a cystectomy- Standard of Care Group: Patients will receive standard of care treatment. Patients will be asked to complete the Demoralization Scale II and Female Sexual Function Index at baseline, 1-month following treatment, 3-months following treatment, 6-months following treatment, and one-year following treatment.
  Interventions: Other: Questionnaires
- Patients receiving a cystectomy - Additional Education Group: Patients will receive additional education with standard of care treatment. Patients will be asked to complete the Demoralization Scale II and Female Sexual Function Index at baseline, 1-month following treatment, 3-months following treatment, 6-months following treatment, and one-year following treatment. Patients will also be asked to complete an attendance diary documenting additional support services utilized. The Attendance Diary will be completed at 1-month following treatment, 3-months following treatment, 6-months following treatment, and one-year following treatment.
  Interventions: Other: Additional Education; Other: Attendance Diary

INTERVENTIONS:
Other: Additional Education — Study-Specific Patient Handouts, Treating-Provider led counseling, Women's Bladder Cancer Support Group, Women's Bladder Cancer Educational Series, and referrals for additional support services
  Groups: Patients not receiving a cystectomy - Additional Education Group; Patients receiving a cystectomy - Additional Education Group
Other: Questionnaires — Female Sexual Function Index, Demoralization Scale-II
  Groups: Patients not receiving a cystectomy - Standard of Care Group; Patients receiving a cystectomy- Standard of Care Group
Other: Attendance Diary — Attendance Diaries for the Women's Bladder Cancer Support Group, Women's Bladder Cancer Educational Series, and additional educational and support services utilized
  Groups: Patients not receiving a cystectomy - Additional Education Group; Patients receiving a cystectomy - Additional Education Group

SUMMARY:
This research is being done to learn more about coping and survivorship of women with bladder cancer, specifically regarding psychosocial distress and sexual dysfunction. This study is a non-therapeutic study and will randomize participants to a standard of care group and education group. Patients in both groups will be asked to complete surveys regarding their mood and sexual function. Patients in the intervention group will be asked to complete attendance diaries regarding educational and support services utilized. Participants' clinical data will also be collected.

DETAILED DESCRIPTION:
The Gender Related Coping and Survivorship Study for Genitourinary Cancers is focused on providing patients with additional education to promote sexual function in female bladder cancer patients with the aim to help decrease demoralization and sexual dysfunction. Patients receiving a cystectomy and patients not receiving a cystectomy will be randomized separately into an additional education or standard of care group. The additional education consists of asking patients to attend the Women and Bladder Cancer Educational Series, Women's Bladder Cancer Support Group meetings, referrals to other support services, receiving supplemental handouts and treating physician led counseling incorporated into standard of care visits. All participants will be asked to complete the Demoralization Scale-II and Female Sexual Function Index at baseline, one-month following treatment, three-months following treatment, six-months following treatment, and one year following treatment. Patients randomized to the additional education group will also be asked to complete an attendance diary one-month following treatment, three-months following treatment, six-months following treatment, and one year following treatment.

ELIGIBILITY:
Inclusion Criteria:

* Females with bladder cancer
* Willing to answer surveys regarding their psychosocial health and sexual health

Exclusion Criteria:

* Not undergoing either active treatment or active surveillance (i.e. patients on hospice care)
* Patients with cognitive impairments
* Women who are pregnant

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Females Diagnosed with Non-Muscle Invasive Bladder Cancer and Muscle Invasive Bladder Cancer
Sampling Method: Probability Sample
Enrollment: 80 (Estimated)
Dates: Start 2023-01-20 (Actual); Primary Completion 2028-09 (Estimated); Study Completion 2029-09 (Estimated)

PRIMARY OUTCOMES:
Use Demoralization Scale-II to assess change in demoralization | Baseline, 1-Month after Treatment, 3-Months after Treatment, 6-Months after Treatment, 1-year after Treatment
  Evaluate educational interventions to improve demoralization in females with bladder cancer. The minimum score is 0 and the maximum score 32. Low scores are defined as 0-3, middle scores are defined between 4-10, and high scores are defined as ≥11.

SECONDARY OUTCOMES:
Use Female Sexual Function Index (FSFI) to assess change in sexual function | Baseline, 1-Month after Treatment, 3-Months after Treatment, 6-Months after Treatment, 1-year after Treatment
  Evaluate if educational interventions improve sexual function in females with bladder cancer. The minimum total score for the FSFI is 2 and the maximum total score is 36. A higher score indicates increased sexual function.
Change in coping as assessed by Demoralization Scale II | Baseline, 1-Month after Treatment, 3-Months after Treatment, 6-Months after Treatment, 1-year after Treatment
  Assess how coping in females with bladder cancer differs by stage of bladder cancer. For the Demoralization Scale II, the minimum score is 0 and the maximum score 32. Low scores are defined as 0-3, middle scores are defined between 4-10, and high scores are defined as ≥11.
Change in coping as assessed by the Female Sexual Function Index (FSFI) | Baseline, 1-Month after Treatment, 3-Months after Treatment, 6-Months after Treatment, 1-year after Treatment
  Assess how coping in females with bladder cancer differs by stage of bladder cancer. The minimum total score for the FSFI is 2 and the maximum total score is 36. A higher score indicates increased sexual function.
Survivorship | Baseline, 1-Month after treatment, 3-Months after Treatment, 6-Months after Treatment, 1-year after Treatment
  Assess survivorship in females with bladder cancer differs by stage of bladder cancer.

CONTACTS AND LOCATIONS:
Overall Officials: Armine Smith, MD, Principal Investigator — Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins
Locations (2):
- United States (2):
  - Sibley Memorial Hospital, Washington D.C., District of Columbia
  - Johns Hopkins Hospital, Baltimore, Maryland

IPD SHARING:
Plan to Share IPD: No